CLINICAL TRIAL: NCT03614611
Title: Canadian Experience With Contiform Intravaginal Device For The Treatment Of Stress Incontinence: Effectiveness And Patient Acceptability
Brief Title: Canadian Experience With Contiform Intravaginal Device For The Treatment Of Stress Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of fund
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Urological Association (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Contiform 2019-4215
Record Dates: First submitted 2018-07-19; First posted 2018-08-03 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Urinary Incontinence, Stress
Keywords: pessaries; Urinary Incontinence/therapy; Patient Satisfaction; Female; Surveys and Questionnaires; Treatment Outcome
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Participants who accept to take part in this study will be assigned to the intervention group. There will be no randomisation or controlled group.
  This study will be taking place in Canada, with the intervention device being approved by Health Canada (Licence No.: 98950, Company ID: 134089, Device identifier: SKU 184)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contiform pessary (Experimental): Enrolled participants will be part of the intervention arm. They will use of the Contiform Intravaginal pessary for the treatment of stress urinary incontinence, for a period of 3 months.
  Interventions: Device: Contiform pessary

INTERVENTIONS:
Device: Contiform pessary — Patients will be asked to use the device for 12 weeks and to become comfortable with self-insertion and self-removal. The device can be worn continuously for 1 month. When placed in the vagina it retains its shape and supports the urethra during episodes of varied intraabdominal pressure. During the assessment test (24 hours pad test), patients will be encouraged to undertake any activity that would normally induce stress leakage.
  The contiform device is approved by Health Canada since 2017-04-10 (Licence No.: 98950, Company ID: 134089, Device identifier: SKU 184)

SUMMARY:
Stress urinary incontinence (SUI) is a highly prevalent condition of involuntary urine leakage associated with coughing, sneezing or exertion. Midurethral slings (MUS) are a safe and efficacious surgical option to treat SUI and is considered the best treatment by recognized organizations. Nevertheless, it remains a surgical intervention exposing patients to risks, possible recurrence and is not recommended to women planning to have more children. Incontinence pessaries offer an alternative to surgery with a similar mechanism of action as MUS. However, there is a paucity of literature on the outcomes of incontinence pessary treatment of SUI, with only two prospective studies have been published on the Uresta pessary and one australian case-series on Contiform pessary.

The objective of the study is to evaluate the effectiveness of the self-positioning Contiform intravaginal pessary used as a conservative method to address stress urinary incontinence in women in order to provide Canadian real-world data.

The 3-month efficacy, adverse events and global patient satisfaction (including comfort and ease of insertion) will be assessed.

It is hypothesized that the Contiform device will be well tolerated by 60-70% of patients, with no serious adverse events. It will cure SUI for about 50% of them.

DETAILED DESCRIPTION:
Patient who will present to the investigator's tertiary urology clinic with the main complaint of stress incontinence will be invited to consider the Contiform device. A total of 50 women will be recruited and followed over 3 months.

The evaluation of enrolled women will include a medical history and physical examination, a urinalysis, a urine culture, three-day voiding diary and post-void residual (PVR). Urodynamic testing will not be required. Kegel assessment will be performed on physical pelvic exam based on the Oxford subjective scale, which ranged from 0 (no palpable contraction) to 5 (very strong contraction). Demographic and baseline characteristics of the participants will be recorded, medical condition and medication.

Patients will be offered the Contiform device and invited to join the study as one treatment option for their stress leak. Patients will be asked to use the device for 12 weeks and to become comfortable with self-insertion and self-removal. All postmenopausal women will be given topical vaginal estrogen therapy before or on the day of starting using the device. No other treatment will be initiated during the trial period.

Once enrolled, patients will be given brief verbal and written instructions on pessary insertion and cleaning, and then allowed to select and insert the pessary themselves at home. They will be provided with a New User Kit which comprises three available sizes (Small, Medium & Large) and a Silicone Removal Strap.

Patient enrolled will have to sign a informed consent form and agree that all information obtained during the research will be kept and treated confidentially within the limits of the law. The results of this study may be published or communicated in other ways; however, no identity or any other identifying information will not be disclosed in any reports or publications. The confidential records and data may be kept up to 10 years.

Patient will have to come to 3 visits. The first one for enrolment and baseline data collection with an urologist, a second visit at 4 weeks with a research nurse assistant and a last one at 3 months with the urologist. On each visit, any adverse event not by the patient of find on physical examination will be note. Test, exam and questionnaire will also be performed (urinalysis and urine culture, to exclude Urinary Tract Infection, residual urine estimation by ultrasonography, a 3-day voiding diary, a 24 hours pad weight test, a vaginal speculum exam performed to look for abrasions or other abnormalities and the completion of questionnaire on quality of like (PGI-I, ICIQ, UDI-6 and a pessary use questionnaire)

Statistical analysis will be performed using the Statistical Package for the Social Sciences (SPSS) (version13, SPSS Inc, Chicago, IL). All data will be described as the median value plus the interquartile range (IQR), as the data will probably not be normally distributed. Wilcoxon's and the Mann-Whitney U tests will be used for paired and unpaired data, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Complain of stress incontinence
* Sufficient manual dexterity to insert and remove the device;
* Ability to speak French or English and understand written informed consent as per local ethical committee approval.

Exclusion Criteria:

* a main complaint of urgency symptoms, bacterial cystitis (symptomatic or proven UTI) at the time of insertion, recent pelvic surgery within the last 3 months, previous pelvic radiotherapy, current pregnancy, failed use of an incontinence pessary, a functional bladder capacity on bladder diary less than 250 mL, prolapse of any vaginal compartment beyond the level of the hymen, post-void residual urine volume greater than 100 mL, hematuria, undiagnosed pelvic or vaginal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The goal of the study is to evaluate the effectiveness of the self-positioning Contiform intravaginal pessary used as a conservative method to address stress urinary incontinence. It can only be use in women.
Enrollment: 39 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the Contiform intravaginal pessary to achievement a change of 50 % or greater reduction in pad weight at 3 months compare to baseline | 3 months
  The primary outcome measure will be the 24-h pad test before and after device placement. In order to determine whether the device is equally effective in mild or more severe leakage, two groups will be analyzed separately. A leakage of <100 g/24h will be categorized as "mild loss" and >100 g/24h will be termed "moderate/severe loss". A weight of less than 2 g will be considered normal. Baseline data will be compare to 3 months to assess change.

SECONDARY OUTCOMES:
Assessment of any new adverse symptoms | 4 weeks and 3 months
  Assessment by a nurse or doctor for any new symptoms reported by the patient. Symptoms could range from a feeling of incomplete emptying, pain/discomfort, urgency, bowel symptoms to hemoserous staining/discharge. Assessment will be taken at the fourth week and the third month visits.
Assessment of device defect | 4 weeks and 3 months
  Assessment by a nurse or doctor for any defects appearing on the device, at the fourth week and the third month visits.
Assessment of augmentation of residual urine volume as an adverse event | 4 weeks and 3 months
  Assessment by a nurse or doctor for the adverse event of augmentation of residual urine volume (mL), measure by bladder scan (ultrasound) after a full miction. Assessment will be taken at the fourth week and the third month visits.
Assessment of vaginal adverse event | 4 weeks and 3 months
  Assessment by a nurse or doctor for any new vaginal adverse event caused by the device, such as vaginal abrasion or other abnormality. Assessment will be done by a speculum vaginal exam at the fourth week and the third month visits.
Patient quality of life and urinary incontinence symptoms as assessed by the ICIQ | 4 weeks and 3 months
  Patients will be asked to complete the International Consultation on Incontinence Questionnaire (ICIQ). The total score is report, with the minimum result being 0 (no symptoms of urinary incontinence) and the maximum being 21 (maximum urinary incontinence as report by this self-taken questionnaire). This questionnaire will be assess at the fourth week and the third month visits.
Patient quality of life and discomfort regarding their urinary incontinence symptoms as assessed by the UDI-6 | 4 weeks and 3 months
  Patients will be asked to complete the urogenital distress inventory (UDI-6) questionnaire. Each item is scored between 0 (no problem) to 3 (bothered greatly). All scores are summed and divided by 6, then multiplied by 33.3 for the scale score. Higher score (100) indicate higher disability. This questionnaire will be assess at the fourth week and the third month visits.
Patient perception of efficacy and their acceptability of the device as assessed by the PGI-I | 4 weeks and 3 months
  Patients will be asked to complete the Patient Global Impression of Improvement (PGI-I). The scale is from 1 to 7, with the highest result being a impression of having a much worse condition with the treatment, and the lowest result (1) is the impression of a very good improvement.This questionnaire will be assess at the fourth week and the third month visits.
Patient acceptability and use of the device, as assessed by the Pessary Use Questionnaire | 4 weeks and 3 months
  Patients will be asked to complete the pessary use questionnaire. The minimum score is 0 and the maximum is 18. The highest result is associated with a better outcome in terms of acceptability and improvement of quality of life. The first 4 questions are using a Likert-type scale (0 to 4), with the maximum associated with a better outcome (improvement or utilisation acceptability), and the last 2 are polar questions. This questionnaire will be assess at the fourth week and the third month visits.

CONTACTS AND LOCATIONS:
Overall Officials: Genevieve Nadeau, MD,MSc,FRCSC, Principal Investigator — CHU de Québec - Université Laval
Locations (1):
- Hopital St-François d'Assise, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen WA, Leek H, Izurieta A, Moore KH. Update: the "Contiform" intravaginal device in four sizes for the treatment of stress incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jun;19(6):757-61. doi: 10.1007/s00192-007-0519-1. PMID 18183342
- [Background] Farrell SA, Baydock S, Amir B, Fanning C. Effectiveness of a new self-positioning pessary for the management of urinary incontinence in women. Am J Obstet Gynecol. 2007 May;196(5):474.e1-8. doi: 10.1016/j.ajog.2006.11.038. PMID 17466709
- [Background] Lovatsis D, Best C, Diamond P. Short-term Uresta efficacy (SURE) study: a randomized controlled trial of the Uresta continence device. Int Urogynecol J. 2017 Jan;28(1):147-150. doi: 10.1007/s00192-016-3090-9. Epub 2016 Jul 20. PMID 27438055
- [Background] Wein AJ, Kavoussi LR, Partin AW, Peters C. Campbell-Walsh urology. 11e ed. Philadelphia, Pennsylvania: Elsevier; 2016